CLINICAL TRIAL: NCT00960973
Title: The Effect of Vitamin K Supplementation on Glucose Metabolism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Chan Soo, Shin, Seoul National University Medical School
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Vitamin K
Record Dates: First submitted 2009-08-16; First posted 2009-08-18 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Diabetes; Prediabetic State
Keywords: vitamin K; beta cell; glucose metabolism; insulin resistance
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State; Insulin Resistance | interventions — menatetrenone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin K (Experimental): Vitamin K supplementation (menatetrenone 30 mg, 3 times a day for 4 weeks)
  Interventions: Drug: Menatetrenone
- Placebo control (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Menatetrenone — Menatetrenone 30 mg, 3 times a day for 4 weeks
  Arms: Vitamin K
Drug: Placebo — Placebo
  Arms: Placebo control

SUMMARY:
The purpose of this study is to test whether vitamin K supplementation has an effect on glucose metabolism in terms of acute beta cell response.

DETAILED DESCRIPTION:
Recently, many studies have reported that vitamin K metabolism is related to glucose metabolism. The suggested mechanisms connecting vitamin K metabolism and glucose metabolism, are inflammation responses and osteocalcin effect on glucose metabolism. Most of the studies have investigated fasting glucose and insulin sensitive index, few have assessed glucose-intake-stimulated responses in regard to vitamin K supplementation. The purpose of this study is to test whether vitamin K supplementation has an effect on glucose metabolism in terms of acute beta cell response using intravenous glucose tolerance test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteer older than 20 years

Exclusion Criteria:

* Subjects with (a history of) diabetes
* Subjects receiving medication related to diabetes or obesity
* Subjects receiving warfarin

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
AIRg (acute insulin response to glucose) using FSIGT (frequently sampled intravenous glucose tolerance test) | 4 weeks later

SECONDARY OUTCOMES:
beta-cell function (FSIGT) | 4 weeks later
disposition index (FSIGT) | 4 weeks later
insulin sensitivity (FSIGT) | 4 weeks later

CONTACTS AND LOCATIONS:
Overall Officials: Chan Soo Shin, MD, PhD, Principal Investigator — Seoul National University Medical School
Locations (1):
- Seoul National University Medical School, Seoul, South Korea